CLINICAL TRIAL: NCT05672940
Title: Investigations of the Effects and Associated Neural Mechanisms of Different Long-term Exercise Interventions on Improving Brain, Cognitive, and Physical Functions in Middle-aged and Older Adults With Metabolic Syndrome
Brief Title: Investigations of the Effects and Associated Neural Mechanisms of Different Exercise in People With Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201912239RINB; MOST 111-2314-B-002-163 - (Other Grant/Funding Number: Ministry of Science and Technology, Taiwan)
Record Dates: First submitted 2022-12-19; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Physical Activity
Keywords: Neuroimage; Training; Aging; Brain; Cardiovascular risks; Metabolic syndrome
MeSH Terms: conditions — Motor Activity; Metabolic Syndrome | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic plus resistance training group (Experimental): Receive three one-hour supervised group sessions weekly for 12 weeks, in which Sections 1 and 3 were AT plus RT sessions, including 5-minute warm-up, 30-minute AT exercises on a bicycle (Comfort 408, Horizon Fitness) or a treadmill (832T, Horizon Fitness), 20-minute RT, and 5-minute cool-down; whereas Section 2 was an AT-only session, including 5-minute warm up, 50-minute aerobic exercises (bicycling or treadmill walking), and 5-minute cool-down.
  Interventions: Behavioral: Aerobic plus resistance training
- Stretching plus breathing training group (Experimental): Receive three one-hour sessions of weekly supervised group training combining Tongtze Gymnastics (童子體操) and breathing exercises for 12 weeks.
  Interventions: Behavioral: Stretching plus breathing training

INTERVENTIONS:
Behavioral: Aerobic plus resistance training — Aerobic plus resistance training
  Arms: Aerobic plus resistance training group
Behavioral: Stretching plus breathing training — Stretching plus breathing training
  Arms: Stretching plus breathing training group

SUMMARY:
Metabolic syndrome (MetS) is a risk for many chronic diseases of middle-aged and older adults. Hence, prevention and treatment of MetS is a crucial global health issue. However, it remains unclear regarding the cognitive effects and associated neural mechanisms of exercise interventions in this population. Therefore, the aims of this three-year project are to compare the effects and neural mechanism of three different types of exercise interventions, on components of MetS, as well as neuropsychological and physical functions in middle-aged and older adults with MetS.

DETAILED DESCRIPTION:
This three-year study is an assessor-blind randomized controlled clinical trial. Another 67 middle-aged and older adults with MetS without regular exercise habits will be recruited and randomly assigned into the combined aerobic and resistance training (AT/RT) or Control (stretching and breathing exercise, ST/BR) group. All participants will undertake three one-hour sessions of exercises for 12 weeks, being supervised . Participants will also wear a wearable device that monitors, records, and provides feedback about their physical activity levels and heart rates during the entire 12 weeks. The outcome measures include participants's components of MetS and performance on neuropsychological and physical tests and structural and functional brain imaging parameters collected at pre-training, and post-training (week 12) tests. The investigators will compare the differences on all of these outcome measures and analyze the relationships between changes in brain structure and functional activation in relationship with other outcome measures in order to understand the neural mechanisms of the training effects and the differences in these mechanisms between the two groups.

Results of this study will provide important scientific evidence and clinical decision bases for determining effective exercise interventions in preventing the progression of MetS, improving neuropsychological and physical functions of MetS, as well as elucidating the neural mechanisms underlying these improvements.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 80 years old
* Literacy
* Diagnosed with MetS based on the International Diabetes Federation (IDF) definition (Alberti et al., 2006) The IDF definition of MetS includes central obesity, determined by waist circumference at the midpoint between the lowest rib and iliac crest being ≧ 90 cm for men and ≧ 80 cm for women, plus at least two of the following conditions- (a) TG ≧ 150 mg/dl or being treated for this lipid abnormality, (b) HDL-C < 40 mg/dl in men, < 50 mg/dl in women, or being treated for this lipid abnormality, (c) systolic blood pressure (SBP) ≧ 130 mmHg, or systolic blood pressure (DBP) ≧ 85 mmHg, or being treated for diagnosed hypertension, and (d) FPG ≧ 100 mg/dl or diagnosed Type II DM).
* Living with a sedentary lifestyle (defined as being engaged in physical activities for less than a total of 90 minutes per week) (Fletcher et al., 1996) in recent one year.

Exclusion Criteria:

* Having any contraindications for fMRI (e.g., claustrophobia and indwelling metals or implanted devices)
* Serious or uncontrolled cardiovascular or pulmonary conditions (e.g., unstable angina, serious cardiac arrhythmias, heart failure, hypertrophic cardiomyopathy, severe aortic or carotid stenosis, pulmonary embolus or infarction, resting SBP ≥ 180 mmHg, or resting DBP ≥ 110 mmHg)
* Severe renal failure (Stages 4 and 5 of chronic kidney diseases (Levin et al., 2013)
* Symptoms or histories of neurological diseases, including transient ischemic attack
* Severe musculoskeletal disorders which would affect their mobility
* Diagnosis of dementia, Montreal Cognitive Assessment (MoCA) (Taiwan version) < 22 (Tsai et al., 2012; Wang et al., 2013), or inability to follow instructions
* Psychiatric disorders (including depression) or Geriatric Depression Scale-short form (GDS-15) score≧8 (Sheikh & Yesavage, 1986)
* Having contraindications for doing exercises (e.g., resting SBP ≥ 180 mmHg, resting DBP ≥ 110 mmHg, FPG ≥ 300 mg/dL, hypoglycemia (plasma glucose ≤ 70 mg/dL) after exercises, or postural hypotension (BP drop ≥ 20 mmHg when changing postures)
* Life expectancy less than six months due to any disease.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of brain functional activation and structure imaging | at baseline, 12 weeks exercise intervention
  Functional Magnetic Resonance Imaging (fMRI) activation patterns and white and gray matter changes of the brain

SECONDARY OUTCOMES:
Neuropsychological test-CANTAB | at baseline, 12 weeks exercise intervention
  Cambridge Neuropsychological Test Automated Battery
Neuropsychological test-AD8 | at baseline, 12 weeks exercise intervention
  Ascertain Dementia-8
Neuropsychological test-MoCA | at baseline, 12 weeks exercise intervention
  Montreal Cognitive Assessment-Taiwan version
Neuropsychological test-CDR | at baseline, 12 weeks exercise intervention
  Clinical Dementia Rating
Neuropsychological test-CTT | at baseline, 12 weeks exercise intervention
  Color Trail Test (in seconds)
Physical test-Muscle strength | at baseline, 12 weeks exercise intervention
  Bilateral grip strength and knee extensor strength (in kilograms)
Physical test-Flexibility | at baseline, 12 weeks exercise intervention
  Chair Sit and Reach Test, The upper extremity and lower extremity/trunk flexibility were measured with the Scratch Test (in centimeters)
Physical test-Balance and mobility | at baseline, 12 weeks exercise intervention
  One-legged Standing (in seconds)
Physical test-Balance and mobility | at baseline, 12 weeks exercise intervention
  Chair Rise Test (in seconds)
Physical test-Balance and mobility | at baseline, 12 weeks exercise intervention
  Four Square Step Test (in seconds)
Physical test-Gait mat | at baseline, 12 weeks exercise intervention
  Gait analysis
Physical test-Heart rate variability | at baseline, 12 weeks exercise intervention
  Heart rate variability
Physical test-Cardiovascular fitness | at baseline, 12 weeks exercise intervention
  Cardiovascular fitness: 6-minute Walk Test
Cardiopulmonary test | at baseline, 12 weeks exercise intervention
  Cycling on the cycle ergometer: Indicate participant's submaximal and maximal cardiovascular fitness level, respectively, and served as references when setting participant's target heart rate for exercise training
Number of participants with Abnormal Laboratory Values | at baseline, 12 weeks exercise intervention
  The following MetS and cardiovascular risk related biomarkers: total cholesterol, triglyceride, HDL, LDL, Fasting plasma glucose, fasting plasma insulin, HbA1c, serum adiponectin level, serum leptin level, and homocysteine

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Fang Tang, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Collage of Public Health, Taipei, Zhongzheng, Taiwan